CLINICAL TRIAL: NCT06747741
Title: Effects of PNF Stretching vs Conventional Physical Therapy on the Symptoms of Restless Leg Syndrome in Elderly Population.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/44
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-10

CONDITIONS: Elderly; Restless Leg Syndrome (RLS); Proprioceptive Neuromuscular Facilitation; Sleep Disturbance
Keywords: Elderly; Restless Leg Syndrome; Sleep Disturbance; PNF stretching; Proprioceptive neuromuscular facilitation
MeSH Terms: conditions — Restless Legs Syndrome; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Stretching technique Group (Experimental): The participants will receive PNF stretching technique of contract-Relax with agonist contraction for 3 days per week on alternate days for the symptoms of RLS in elderly population.
  Interventions: Procedure: PNF stretching(Contract relax with agonist contraction)
- Conventional physical therapy Group (Active Comparator): The participants will receive Conventional physical therapy including calf stretchinf and strenthening exercises, 3 days per week on alternative days for the symptoms of RLS in elder population.
  Interventions: Procedure: Conventional physical therapy

INTERVENTIONS:
Procedure: PNF stretching(Contract relax with agonist contraction) — 1.Passively dorsiflex the patient's foot then ask to perform active planterflexion against resistance and hold for 7-10 sec then ask patient to perform dorsiflexion to the maximum available range.
  Arms: PNF Stretching technique Group
Procedure: Conventional physical therapy — Static Stretching:(Seated Calf Stretch With a Resistance Band)
  1. Sit on the floor with your legs extended.
  2. Loop a resistance band around one foot, holding both sides of it with your hands.
  3. Gently pull your toes toward your shin until you feel the stretch in your calf.Repeat on the other side.
  Isometric Calf Raise:
  1. Stand with feet shoulder-width apart and arms at sides.
  2. Engage your abs for stability and roll up onto the balls of your feet, lifting both heels off the floor.
  3. Hold for 5 seconds, then return to the starting position. Frequency : 5 reps with 5-7Sec hold,3 days per week for 4 weeks (alternatively)
  Arms: Conventional physical therapy Group

SUMMARY:
Restless leg Syndrome (RLS) is a common condition in the elderly population,characterized byan uncontrollable urge to move the leg,often occuring in the evening or at night,which can significantly disturb sleep and daily activities(ADL).

Although various type of stretchings found to be effective on the symptoms of RLS,no study has specifically compared the effects of Proprioceptive Neuromuscular Facilitation stretching technique versus conventional physical therapy on the symptoms of RLS and related sleep disturbances.This study aims to fill this gap by evaluating the effectiveness of PNF stretching compared to conventional physical therapy,on the symptoms of RLS in elderly population.

DETAILED DESCRIPTION:
OBJECTIVES:

Objectives of this study are:

1. To determine the effect of PNF stretching VS conventional physical therapy on the symptoms of Restless leg syndrome in elder population.
2. To determine the effect of PNF stretching VS conventional physical therapy on sleep disturbance related to restless leg syndrome in elder population.

HYPOTHESIS:

Alternate Hypothesis:

1. There is statistically significant difference between the effect of PNF stretching VS Conventional physical therapy on the symptoms of Restless leg syndrome in elder population.
2. There is statistically significant difference between the effect of PNF stretching VS conventional physical therapy on the sleep disturbance related to restless leg syndrome in elder population.

Null Hypothesis:

1. There is no statistically significant difference between the effect of PNF stretching VS conventional physical therapy on the symptoms of Restless leg syndrome in elder population.
2. There is no statistically significant difference between the effect of PNF stretching VS conventional physical therapy on sleep disturbance related to restless leg syndrome in elder population.

Study Design: Randomized Controlled Trial

Clinical setting: Fauji foundation Hospital(Rehab Depart) Islamabad Healing Center. Study Duration: 1year

SELECTION CRITERIA:

Inclusion Criteria:

1. Age 60 and above.
2. Both male and female.
3. Must fulfil the diagnostic criteria of primary restless leg syndrome.

Exclusion Criteria:

1.A history or underlying disease that would contribute to the syptoms of RLS.

Sampling Technique:Non probability purposive samping.

Data will be collected on demographics and general information. Data will be coollected using International Restless leg syndrome rating scale,Post-sleep questionnaire.

Experimental Group:This group will receive PNF stretching technique of Hold-relax with agonist contraction,outcome will measure before and after the treatment of 4 weeks.

Control Group:This group will receive conventional physical therapy,Outcome will measure before and after 4 weeks of treatment.

Data will be analyze through SPSS21 and data will be analyzed based on study design choosen that is Randomize control study with in the community.

The printed questionnaire will be provided to the patients after obtaining written consent and providing adequate information regarding the study,after which the data will be presented in the form of graphs or tables.

Significance of the study:

Although PNF stretching proves to be more effective in reducing pain increasing ROM and flexibility,but there is limited documentation about its effect on RLS.

This study aims to uncover and augument the treatment strategies that can wield even more favourable results in elder population dealing with Restless leg syndrome and also sleep disturbance related to it.

So it will aid therapist in choosing right technique saving their time and patient's investment.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and above.
* Male & Females both.
* must fulfill the diagnostic criteria of primary RLS.

Exclusion Criteria:

* A history or underlying disease that would contribute to the symptoms of RLS.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Severity of restless leg syndrome symptoms | 4 weeks
  International Restless leg syndrome rating scale is 10 item Questionnaire,each question has 0(None) to 4(very severe) grading.Total score is 40,Mild(1-10),Moderate(11-20),Severe(21-30),Very severe(31-40).Participant will be assessed through this scoring system for the severity of RLS symptoms.
Sleep disturbance related to RLS | 4 weeks
  5 Item questionnaire related to quality of sleep.Higher score indicate higher sleep disturbance.quality of sleep of participant will be assess through this questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan